CLINICAL TRIAL: NCT04637243
Title: Evaluation of Outcomes From Treatment of Benign or Malignant Liver and Bile Duct Diseases
Brief Title: Outcomes From Treatment Liver and Bile Duct Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 035.HPB.2018.R
Record Dates: First submitted 2019-09-12; First posted 2020-11-19 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-03

CONDITIONS: Benign or Malignant Liver and Bile Duct Disease
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment of Benign or Malignant Liver and Bile Duct Diseases — Available treatment of Benign or Malignant Liver and Bile Duct Diseases

SUMMARY:
It is reported in the literature that the treatment of any liver and bile duct disease process, whether benign or malignant, continues to be a huge challenge. For example, patients with adenocarcinoma continue to be diagnosed at an advanced stage with medical and surgical options that are improving in terms of outcome measurements but with much more room for improvement. Our goal is to continue to review our treatment outcomes to further improve overall survival, overall symptom control, mortality and morbidity.

The main aim of this study is to evaluate and compare the outcomes from our multiple treatments of benign or malignant liver and bile duct diseases.

DETAILED DESCRIPTION:
The study will be a retrospective chart review of patients who have been diagnosed with benign or malignant liver and bile duct disease under the practices of Rohan Jeyarajah, M.D., Houssam Osman, M.D., F.A.C.S., Edward Cho, M.D., Sc.M at Methodist Health System Hospital in Richardson, T.X. We plan to conduct an analysis of patients meeting the inclusion criteria form 2005 to present (up to the day before this study receives IRB approval). Charts will also be reviewed by the PI. Sub-I, Fellows, Office Staff, Clinical Research Coordinator who are delegated to do so by the PI. Data will be obtained from a national database. Data will be analyzed primarily by the study conductors.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed and treated for liver and bile duct disease benign or malignant from 2005 to present (up to the day before this study receives IRB approval)
* Age > 18 years

Exclusion Criteria:

* Patients that are not diagnosed with or treated for liver and bile duct disease
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been diagnosed with benign or malignant liver and bile duct disease under the practices of Rohan Jeyarajah, M.D., Houssam Osman, M.D., F.A.C.S., Edward Cho, M.D., Sc.M at Methodist Health System Hospital in Richardson, T.X.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality from Treatment of Benign or Malignant Liver and Bile Duct Diseases | 2005 to 2019
  Mortality
Morbidity from Treatment of Benign or Malignant Liver and Bile Duct Diseases | 2005 to 2019
  Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Dhiresh Jeyarajah, M.D., Principal Investigator — Trinity Surgical Consultants, Methodist Richardson Medical Center
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No